CLINICAL TRIAL: NCT03542110
Title: Effect of Alirocumab on Saphenous Vein Graft Atherosclerosis: The Alirocumab for Stopping Atherosclerosis Progression in Saphenous Vein Grafts (ASAP-SVG) Pilot Trial
Brief Title: The Alirocumab for Stopping Atherosclerosis Progression in Saphenous Vein Grafts (ASAP-SVG) Pilot Trial
Acronym: ASAP-SVG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawal of medication and funding support by Sponsor
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASAP-SVG, QR#32711/1
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Saphenous Vein Graft Atherosclerosis
MeSH Terms: interventions — alirocumab; Injections, Subcutaneous; Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alirocumab 150 MG/ML subcutaneous injection (Active Comparator): Alirocumab 150 mg subcutaneously every 2 weeks
  Interventions: Drug: Alirocumab 150 MG/ML subcutaneous injection
- Matching Placebo subcutaneous injection (Placebo Comparator): Matching placebo subcutaneously every 2 weeks
  Interventions: Drug: Matching Placebo subcutaneous injection

INTERVENTIONS:
Drug: Alirocumab 150 MG/ML subcutaneous injection — Single-dose, pre-filled, disposable, subcutaneous injection pen
  Other Names: Praluent, Study Drug
  Arms: Alirocumab 150 MG/ML subcutaneous injection
Drug: Matching Placebo subcutaneous injection — Single-dose, pre-filled, disposable, subcutaneous injection pen
  Other Names: Placebo, Study Drug
  Arms: Matching Placebo subcutaneous injection

SUMMARY:
This is a phase IV, multi-center, double-blind, randomized, placebo- controlled study evaluating the effect of alirocumab on SVG atherosclerotic disease burden, as assessed by IVUS at baseline and following 78 weeks of treatment in subjects with at least one intermediate SVG lesion receiving optimal statin therapy. Subjects will be randomized 1:1 into 2 treatment groups: alirocumab 150 mg subcutaneously every 2 weeks or placebo subcutaneously every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater.
2. Willing and able to give informed consent. The patients must be able to comply with study procedures and follow-up.
3. Undergoing clinically-indicated coronary and SVG angiography.
4. Have at least one target saphenous vein graft with an intermediate SVG lesion (defined as a lesion with 30-60% angiographic diameter stenosis) amenable to examination with IVUS. The SVG should have no thrombus or ulceration and should not be considered responsible for the patient's clinical presentation and referral for angiography.
5. Receiving optimal statin therapy defined as use of a high intensity statin (atorvastatin 40-80 mg daily or rosuvastatin 20-40 mg daily), any statin therapy with achieved LDL-C level <70mg/dL, or maximally-tolerated statin dose for patients who are statin intolerant statin.

Exclusion Criteria:

1. Positive pregnancy test or breast-feeding.
2. Coexisting conditions that limit life expectancy to less than 18 months or that could affect a patient's compliance with the protocol.
3. Estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2.
4. Severe peripheral arterial disease limiting vascular access.
5. History of allergic reaction to iodine-based contrast agents that cannot be premedicated.
6. Known hypersensitivity to alirocumab.
7. Any prior use of proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Nominal change in intermediate SVG lesion percent atheroma volume (PAV) from baseline to 78 weeks post randomization, as assessed by intravascular ultrasonography (IVUS). | 78 weeks
  To evaluate the effect of alirocumab on the change in burden of saphenous vein graft (SVG) atherosclerosis as measured by percent atheroma volume (PAV) in patients with intermediate SVG lesions who are undergoing clinically-indicated coronary angiography and are receiving optimal statin therapy.

SECONDARY OUTCOMES:
Nominal change in TAV and normalized TAV of an intermediate SVG lesion from baseline to 78 weeks | 78 weeks
  evaluate the effect of alirocumab on the change in total and normalized total atheroma volume (TAV) of an intermediate SVG lesion
Angiographic failure of target SVG lesion from baseline to 78 weeks. | 78 weeks
  To evaluate the effect of alirocumab on the incidence of angiographic failure of an intermediate target SVG lesion.
Incidence of target SVG failure and major adverse cardiac events. | Randomization to 80 weeks
  To evaluate the effect of alirocumab on the incidence of target SVG failure (defined as the composite of death, myocardial infarction, and target lesion revascularization) and the incidence of major adverse cardiac events (MACE, defined as the composite of death, acute coronary syndrome, or coronary revascularization) during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Study Chair — Minneapolis Heart Institute and Foundation/ Abbott Northwestern Hospital-Allina Health
Locations (4):
- United States (4):
  - San Francisco VA Medical Center, San Francisco, California
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Minneapolis Heart Institute/ Abbott North Western Hospital-Allina Health, Minneapolis, Minnesota
  - Dallas VA Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domanski MJ, Borkowf CB, Campeau L, Knatterud GL, White C, Hoogwerf B, Rosenberg Y, Geller NL. Prognostic factors for atherosclerosis progression in saphenous vein grafts: the postcoronary artery bypass graft (Post-CABG) trial. Post-CABG Trial Investigators. J Am Coll Cardiol. 2000 Nov 15;36(6):1877-83. doi: 10.1016/s0735-1097(00)00973-6. PMID 11092659
- [Background] DeFrances CJ, Lucas CA, Buie VC, Golosinskiy A. 2006 National Hospital Discharge Survey. Natl Health Stat Report. 2008 Jul 30;(5):1-20. PMID 18841653
- [Background] Alexander JH, Hafley G, Harrington RA, Peterson ED, Ferguson TB Jr, Lorenz TJ, Goyal A, Gibson M, Mack MJ, Gennevois D, Califf RM, Kouchoukos NT; PREVENT IV Investigators. Efficacy and safety of edifoligide, an E2F transcription factor decoy, for prevention of vein graft failure following coronary artery bypass graft surgery: PREVENT IV: a randomized controlled trial. JAMA. 2005 Nov 16;294(19):2446-54. doi: 10.1001/jama.294.19.2446. PMID 16287955
- [Background] Sabik JF 3rd. Understanding saphenous vein graft patency. Circulation. 2011 Jul 19;124(3):273-5. doi: 10.1161/CIRCULATIONAHA.111.039842. No abstract available. PMID 21768550
- [Background] Shroyer AL, Grover FL, Hattler B, Collins JF, McDonald GO, Kozora E, Lucke JC, Baltz JH, Novitzky D; Veterans Affairs Randomized On/Off Bypass (ROOBY) Study Group. On-pump versus off-pump coronary-artery bypass surgery. N Engl J Med. 2009 Nov 5;361(19):1827-37. doi: 10.1056/NEJMoa0902905. PMID 19890125
- [Background] Goldman S, Zadina K, Moritz T, Ovitt T, Sethi G, Copeland JG, Thottapurathu L, Krasnicka B, Ellis N, Anderson RJ, Henderson W; VA Cooperative Study Group #207/297/364. Long-term patency of saphenous vein and left internal mammary artery grafts after coronary artery bypass surgery: results from a Department of Veterans Affairs Cooperative Study. J Am Coll Cardiol. 2004 Dec 7;44(11):2149-56. doi: 10.1016/j.jacc.2004.08.064. PMID 15582312
- [Background] Fitzgibbon GM, Kafka HP, Leach AJ, Keon WJ, Hooper GD, Burton JR. Coronary bypass graft fate and patient outcome: angiographic follow-up of 5,065 grafts related to survival and reoperation in 1,388 patients during 25 years. J Am Coll Cardiol. 1996 Sep;28(3):616-26. doi: 10.1016/0735-1097(96)00206-9. PMID 8772748
- [Background] Lichtenwalter C, de Lemos JA, Roesle M, Obel O, Holper EM, Haagen D, Saeed B, Iturbe JM, Shunk K, Bissett JK, Sachdeva R, Voudris VV, Karyofillis P, Kar B, Rossen J, Fasseas P, Berger P, Banerjee S, Brilakis ES. Clinical presentation and angiographic characteristics of saphenous vein graft failure after stenting: insights from the SOS (stenting of saphenous vein grafts) trial. JACC Cardiovasc Interv. 2009 Sep;2(9):855-60. doi: 10.1016/j.jcin.2009.06.014. PMID 19778774
- [Background] Brilakis ES, Lee M, Mehilli J, Marmagkiolis K, Rodes-Cabau J, Sachdeva R, Kotsia A, Christopoulos G, Rangan BV, Mohammed A, Banerjee S. Saphenous vein graft interventions. Curr Treat Options Cardiovasc Med. 2014 May;16(5):301. doi: 10.1007/s11936-014-0301-x. PMID 24643432
- [Background] Ellis SG, Brener SJ, DeLuca S, Tuzcu EM, Raymond RE, Whitlow PL, Topol EJ. Late myocardial ischemic events after saphenous vein graft intervention--importance of initially "nonsignificant" vein graft lesions. Am J Cardiol. 1997 Jun 1;79(11):1460-4. doi: 10.1016/s0002-9149(97)00171-9. PMID 9185633
- [Background] Knatterud GL, White C, Geller NL, Campeau L, Forman SA, Domanski M, Forrester JS, Gobel FL, Herd JA, Hickey A, Hoogwerf BJ, Hunninghake DB, Terrin ML, Rosenberg Y. Angiographic changes in saphenous vein grafts are predictors of clinical outcomes. Am Heart J. 2003 Feb;145(2):262-9. doi: 10.1067/mhj.2003.113. PMID 12595843
- [Background] Rodes-Cabau J, Facta A, Larose E, DeLarochelliere R, Dery JP, Nguyen CM, Roy L, Proulx G, Gleeton O, Barbeau G, Noel B, Rouleau J, Boudreault JR, Bertrand OF. Predictors of aorto-saphenous vein bypass narrowing late after coronary artery bypass grafting. Am J Cardiol. 2007 Aug 15;100(4):640-5. doi: 10.1016/j.amjcard.2007.03.080. Epub 2007 Jun 27. PMID 17697821
- [Background] Rodes-Cabau J, Bertrand OF, Larose E, Dery JP, Rinfret S, Bagur R, Proulx G, Nguyen CM, Cote M, Landcop MC, Boudreault JR, Rouleau J, Roy L, Gleeton O, Barbeau G, Noel B, Courtis J, Dagenais GR, Despres JP, DeLarochelliere R. Comparison of plaque sealing with paclitaxel-eluting stents versus medical therapy for the treatment of moderate nonsignificant saphenous vein graft lesions: the moderate vein graft lesion stenting with the taxus stent and intravascular ultrasound (VELETI) pilot trial. Circulation. 2009 Nov 17;120(20):1978-86. doi: 10.1161/CIRCULATIONAHA.109.874057. Epub 2009 Nov 2. PMID 19884468
- [Background] Rodes-Cabau J, Bertrand OF, Larose E, Dery JP, Rinfret S, Urena M, Jerez M, Nombela-Franco L, Ribeiro HB, Allende R, Proulx G, Nguyen CM, Boudreault JR, Rouleau J, Roy L, Gleeton O, Barbeau G, Noel B, Cote M, Despres JP, Dagenais GR, DeLarochelliere R. Five-year follow-up of the plaque sealing with paclitaxel-eluting stents vs medical therapy for the treatment of intermediate nonobstructive saphenous vein graft lesions (VELETI) trial. Can J Cardiol. 2014 Jan;30(1):138-45. doi: 10.1016/j.cjca.2013.11.002. Epub 2013 Nov 6. PMID 24365196
- [Background] Kotsia AP, Rangan BV, Christopoulos G, Coleman A, Roesle M, Cipher D, de Lemos JA, McGuire DK, Packer M, Banerjee S, Brilakis ES. Effect of Extended-Release Niacin on Saphenous Vein Graft Atherosclerosis: Insights from the Atherosclerosis Lesion Progression Intervention Using Niacin Extended Release in Saphenous Vein Grafts (ALPINE-SVG) Pilot Trial. J Invasive Cardiol. 2015 Oct;27(10):E204-10. PMID 26429851
- [Background] Brilakis ES, Edson R, Bhatt DL, Goldman S, Holmes DR Jr, Rao SV, Shunk K, Rangan BV, Mavromatis K, Ramanathan K, Bavry AA, Garcia S, Latif F, Armstrong E, Jneid H, Conner TA, Wagner T, Karacsonyi J, Uyeda L, Ventura B, Alsleben A, Lu Y, Shih MC, Banerjee S; DIVA Trial Investigators. Drug-eluting stents versus bare-metal stents in saphenous vein grafts: a double-blind, randomised trial. Lancet. 2018 May 19;391(10134):1997-2007. doi: 10.1016/S0140-6736(18)30801-8. Epub 2018 May 11. PMID 29759512